CLINICAL TRIAL: NCT03040479
Title: A Phase I, Multicenter, Open-Label, Parallel-Group, Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetic Single Dose Study of Oral Lasmiditan in Participants With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Algorithme Pharma Inc (Industry); CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16881; CUD-P9-453 (Other: Algorithme Pharma); H8H-CD-LAHF (Other: Eli Lilly and Company); COL MIG-114 (Other: CoLucid Pharmaceuticals)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2018-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, non-randomized, parallel-group, single dose study.
  This study will enroll up to 24 participants and will include 2 hepatic impaired participant groups and one group of control participants with normal hepatic function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Experimental): lasmiditan 200 mg single dose
  Interventions: Drug: lasmiditan 200 mg
- Moderate hepatic impairment (Experimental): lasmiditan 200 mg single dose
  Interventions: Drug: lasmiditan 200 mg
- Healthy participants (Experimental): lasmiditan 200 mg single dose
  Interventions: Drug: lasmiditan 200 mg

INTERVENTIONS:
Drug: lasmiditan 200 mg — single dose
  Other Names: LY573144

SUMMARY:
This is a multicenter, open-label, non-randomized, parallel-group, single dose study. This study will enroll up to 24 participants and will include 2 hepatic impaired participant groups and one group of control participants with normal hepatic function.

DETAILED DESCRIPTION:
This study will enroll up to 24 participants and will include 2 hepatic impaired participant groups and one group of control participants with normal hepatic function. Approximately four participants with mild hepatic impairment will be enrolled first (Group 1). To ensure participant safety, following dosing of these first four participants, a safety meeting will take place to review the safety data prior to dosing additional participants. After safety and pharmacokinetic (PK) results from the first four participants have been reviewed, an additional four participants with mild hepatic impairment (remainder of Group 1) will be enrolled concurrently with the moderate hepatic impairment group (Group 2). Thereafter, matched participants with normal hepatic function (Group 3) will be enrolled. All participants will participate in one treatment period and will receive a single dose of lasmiditan in the fasting state.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Availability for the entire study period
* Motivated participant and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
* Male or female participants
* A female participant of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the drug administration, during the study and for at least 60 days after the dose.
* A male participant with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be unable to procreate, or agrees to use an accepted contraceptive regimens from first drug administration until 3 months after the drug administration.
* A male participant agrees to refrain from sperm donation from drug administration until 90 days after the drug administration
* Participant aged of at least 18 years
* Participant with a body mass index (BMI) greater than or equal to (≥1) 8.5 kilogram per square meter (kg/m²)
* Light-, non- or ex-smokers
* Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF)

Participants with Normal Hepatic Function:

* Clinical laboratory values within the laboratory's stated normal range; if not within this range, these must be without any clinical significance
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, endocrinology, electrocardiogram [ECG], and urinalysis)
* Must match by gender, as well as to the pooled mean values for age (± 10 years) and weight (± 20%) of participants with hepatic impairment

Hepatic Impaired Participants:

* Considered clinically stable in the opinion of the Investigator
* Presence of mild hepatic impairment (Child-Pugh Class A: 5-6 points) or moderate hepatic impairment (Child-Pugh Class B: 7-9 points) at screening

Exclusion Criteria:

All Participants:

* Females who are pregnant or are lactating
* History of significant hypersensitivity to lasmiditan or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Participant is at imminent risk of suicide (positive response to question 4 or 5 on the Columbia- Suicide Severity Rating Scale [C-SSRS]) or had a suicide attempt within 6 months prior to screening
* Presence or history of any disorder (including Parkinson disease) that could interfere with completion of the study based on the opinion of the Principal Investigator
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive results to human immunodeficiency virus antibody/antigen (HIV Ag/Ab) Combo tests (and HIV I & II screen at Orlando Clinical Research Center site)
* Females who are pregnant according to a positive pregnancy test
* Participants who took lasmiditan in the previous 28 days before Day 1 of this study
* Participants who took an Investigational Product (in another clinical trial) in the previous 28 days before day 1 of this study
* Participants who have already participated in this clinical study
* Donation of 500 milliliters (mL) or more of blood in the previous 56 days before day 1 of this study

Participants with Normal Hepatic Function:

* Seated pulse rate less than or equal 50 Beats per Minute (bpm) or more than 100 bpm at screening
* Seated blood pressure below 90/60 millimeters of mercury (mmHg) or higher than 140/90 mmHg at screening
* Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of out-of-range cardiac interval (PR < 110 milliseconds [msec], PR > 220 msec, QRS < 60 msec, QRS >119 msec and QTc > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Positive screening of alcohol and/or drugs of abuse
* Positive results to Hepatitis B surface Antigen (HBsAG [B] [hepatitis B]) or Hepatitis C Virus (HCV [C]) tests
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
* Participants who donated 50 mL or more of blood in the previous 28 days before day 1 of this study

Hepatic Impaired Participants:

* Seated pulse rate less than 40 bpm or more than 110 bpm at screening
* Seated blood pressure below 90/50 mmHg or higher than 170/100 mmHg at screening
* History of hepatic transplant
* Acute exacerbation of hepatic disease within 14 days of study drug administration
* History or presence, in the opinion of the Investigator, of significant clinically unstable respiratory, cardiovascular, pulmonary, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Have poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c >10%
* Evidence of hepatocellular carcinoma present or acute hepatic disease from infection or drug toxicity at the time of screening
* Presence of severe encephalopathy
* Presence of surgically-created or transjugular intrahepatic portal systemic shunts
* History of any major surgery within 6 months before Day 1
* History of bariatric surgery or any other gastrointestinal surgery that may induce malabsorption
* Estimated creatinine clearance by Cockcroft-Gault equation < 40 mL/min/1.73 m² at screening
* Presence of clinically significant physical, laboratory, or ECG finding that, in the opinion of the Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results
* Participants with acute, unstable, or untreated significant medical conditions.
* Positive screening of alcohol and/or drugs of abuse unless results can be explained by a prescription medication
* Participants who donated 100 mL or more of blood in the previous 28 days before day 1 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - NOCCR, Knoxville, Kentucky
- Altasciences Company Inc./Algorithme Pharma, Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male and female adult participants with normal hepatic function, mild and moderate hepatic impairment participated in the study. All participants participated in one treatment period and received a single dose of lasmiditan in the fasting state.Participants confined to the clinic 10 hours prior to dosing until 36 hours after drug administration.
Groups:
- Mild Hepatic Impairment; Moderate Hepatic Impairment; Healthy Participants: Participants received lasmiditan 200 mg single oral dose in the fasting state.
Period: Overall Study
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Started | 8 | 8 | 8
Received at Least 1 Dose of Study Drug | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.2) | 59.1 (7.3) | 58.0 (6.5) | 57.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 2 | 8
  Male | 3 | 7 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 7 | 7 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 8 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 8 | 8
  United States | 8 | 8 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nanograms per milliliter (ng/mL) | 261 (51) | 294 (47) | 220 (25)

2. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time of maximum observed plasma concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hours (hr) | 2.00 [0.75 to 3.00] | 1.38 [0.75 to 2.00] | 2.52 [1.75 to 4.00]

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Tlast (AUC[0-tlast])
Description: Cumulative area under the plasma concentration time curve calculated from 0 to TLQC using the linear trapezoidal method, where TLQC represents time of last observed quantifiable plasma concentration.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nanogram*hour per milliliter (ng*h/mL) | 1750 (38) | 2080 (58) | 1590 (31)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf])
Description: Area under the plasma concentration time curve extrapolated to infinity, calculated as AUC(0-tlast) + CLQC/λZ, where CLQC is the measured concentration at time TLQC Apparent elimination rate constant and λz is the estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL | 1790 (38) | 2170 (59) | 1610 (30)

5. Primary Outcome: Pharmacokinetics: Apparent Elimination Rate Constant (λZ)
Description: Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
1/hour (1/h) | 0.121 (31) | 0.089 (14) | 0.136 (9)

6. Primary Outcome: Pharmacokinetics: Terminal Elimination Half-life (T1/2)
Description: Terminal elimination half-life, calculated as ln(2)/λZ.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable lasmiditan PK data.
Measure: Geometric Mean (Full Range); unit: hours (hr)
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hours (hr) | 5.74 [3.57 to 7.95] | 7.82 [6.58 to 9.54] | 5.09 [4.56 to 5.72]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety assessed from time of consent through end of study (up to 35 days). A summary of all reported serious adverse events (SAE) and other adverse events regardless of causality are provided in the Adverse Events module of this record.
Time Frame: Up To 35 days
Population: All enrolled participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
Participants
  AEs | 3 | 2 | 3
  SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 35 days
Description: All enrolled participants who received at least one dose of the study drug.
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Healthy Participants (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2016-01-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03040479/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03040479/SAP_001.pdf